CLINICAL TRIAL: NCT01297777
Title: Imatinib Mesylate Therapy in Systemic Mastocytosis Patients Lacking KIT Mutations
Brief Title: Imatinib in KIT-negative Systemic Mastocytosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Virgen de la Salud (Other)
Responsible Party: Principal Investigator, LUIS ESCRIBANO, Director Instituto de Estudios de Mastocitosis de Castilla La Mancha, Hospital Virgen de la Salud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2010-019189-94
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Mastocytosis
Keywords: Mast cell; Mastocytosis; Mast cell disease
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis; Mast Cell Activation Disorders | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib mesylate (Experimental): Imatinib mesylate 300 or 400 mg daily for 12 months.
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — * In patients without B or C findings and without biological progression: 300 mg/24 h p.o during one year or until progression/unacceptable toxicity.
  * In patients with B or C findings or biological progression: 300 mg/24 h p.o for two weeks and then 400 mg/24 h p.o for a total of one year of therapy, or until progression/unacceptable toxicity.
  Other Names: Gleevec; STI571

SUMMARY:
The aim of this study is to evaluate the efficacy in terms of clinical and biological response rates of Imatinib Mesylate therapy in patients with systemic mastocytosis lacking KIT mutations.

DETAILED DESCRIPTION:
In vitro studies have proven that imatinib inhibits wild type Kit (wtKit) and suppresses proliferation of the HMC-1V560G cell line, while it is ineffective on inhibiting the growth of HMC-1V560G, D816V cells. Apart from wtKit, Kit molecules carrying mutations in the extracellular, transmembrane and juxtamembrane domains, such as V560G, F522C and K509I, remain sensitive to imatinib. In contrast, several experiments have provided compelling evidence regarding the resistance against the growth-inhibitory effects of imatinib on cells carrying the D816V KIT mutation. As a consequence, sensitive and specific methods should be used in order to avoid "false" KIT mutation-negative cases and, for that purpose, mainly in cases with low bone marrow mast cell numbers, mutational studies should be performed using highly purified bone marrow mast cells by means of Facs sorting systems better than whole bone marrow, unsorted mononuclear cell fraction or mononuclear cell fraction pre-enriched using magnetic beads conjugated with anti-CD25 monoclonal antibody. In the present study mutational studies were performed in all cases in purified bone marrow mast cells (purity > 97%) using a FACSaria system (Becton-Dickinson Biosciences) as previously described.

Patients without B or C findings according to the World Health Organization, and without features of biological progression of the disease receive oral Imatinib Mesylate 300 mg daily for up to 12 months or until clinical progression/unacceptable toxicity. Patients with B or C findings or biological progression initially receive oral Imatinib Mesylate 300 mg daily for two weeks; then, dose is increased up to 400 mg/day except in patients who develop hematological or any other dose-limiting toxicity.

Biological progression is defined as the presence of at least one of the following features: i) increased serum tryptase levels > 200 ng/mL, ii) diffuse bone sclerosis, iii) patchy sclerosis with osteolysis and increased risk of bone fracture or significant bone pain, and, iv) organomegalies or lymph node enlargement due to mastocytosis.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years.
* Diagnosis of systemic mastocytosis in the absence of c-kit mutation.
* ECOG ≤ 3.
* Signed informed consent.

Exclusion Criteria:

* Previous therapy with a tyrosin kinase inhibitor.
* Positive antibodies against HIV or active viral hepatitis.
* Impaired liver function (total bilirubin ≥ 2.0 mg/dl, AST or ALT > 3 x upper limit of normal).
* Impaired renal function (≥ 2.0 mg/dL).
* Grade III-IV cytopenias not related to mastocytosis.
* Severe cardiopathy (grade III/IV of NYHA, or left ventricular ejection fraction < 50%).
* Pregnancy or breastfeeding.
* Female patients who do not use contraceptive methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Imatinib Mesylate on the grade of bone marrow mast cells infiltration. | 6 months
  The grade of bone marrow infiltration is evaluated before and after 6 months of therapy by bone marrow histology and cytology, and flow cytometry performed on highly-purified bone marrow mast cells from patients with B or C findings
To evaluate the effect of Imatinib Mesylate on the grade of bone marrow mast cells infiltration. | 12 months
  The grade of bone marrow infiltration is evaluated before and after 6 months of therapy by bone marrow histology and cytology, and flow cytometry performed on highly-purified bone marrow mast cells from patients without B or C findings, and from those with B or C findings who show response at the intermediate check-point (after 6 months of therapy)

SECONDARY OUTCOMES:
To evaluate the effect of Imatinib Mesylate on mastocytosis skin lesions. | 12 months
  Skin lesions are evaluated before and after therapy by macroscopic examination and skin biopsy.
To evaluate the effect of Imatinib Mesylate on mastocytosis mast-cell related symptoms. | 12 months
  Clinical symptoms such as pruritus, flushing, gastrointestinal symptoms and anaphylaxis are assessed before and after therapy using a clinical questionnaire that includes the type, frequency and severity of each symptom.
To evaluate the effect of Imatinib Mesylate on mastocytosis-related megalies. | 12 months
  Organomegalies and adenomegalies are assessed before and after therapy by abdominal ultrasound.
To evaluate the effect of Imatinib Mesylate on mastocytosis-related bone alterations. | 12 months
  Bone alterations are assessed before and after therapy by X-ray survey.
To investigate changes after Imatinib Mesilate therapy in mast cell clonality. | 12 months
  Genetic abnormalities are assessed before and after therapy by sequencyng analysis of the c-kit gene and the HUMARA assay.
To determine the effect of Imatinib Mesylate therapy on serum tryptase levels. | 12 months
  Serum tryptase is measured before and after therapy.
To determine the effect of Imatinib Mesylate therapy in the psychological impact of the disease and the quality of life. | 12 months
  The psychological impact of the disease and the quality of life of patients are evaluated before and after therapy by the Dermatology Life Quality Index.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Escribano, MD, PhD, Principal Investigator — Instituto de Estudios de Mastocitosis de Castilla La Mancha
Locations (1):
- Instituto de Estudios de Mastocitosis de Castilla La Mancha; Hospital Virgen del Valle, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zermati Y, De Sepulveda P, Feger F, Letard S, Kersual J, Casteran N, Gorochov G, Dy M, Ribadeau Dumas A, Dorgham K, Parizot C, Bieche Y, Vidaud M, Lortholary O, Arock M, Hermine O, Dubreuil P. Effect of tyrosine kinase inhibitor STI571 on the kinase activity of wild-type and various mutated c-kit receptors found in mast cell neoplasms. Oncogene. 2003 Feb 6;22(5):660-4. doi: 10.1038/sj.onc.1206120. PMID 12569358
- [Background] Akin C, Brockow K, D'Ambrosio C, Kirshenbaum AS, Ma Y, Longley BJ, Metcalfe DD. Effects of tyrosine kinase inhibitor STI571 on human mast cells bearing wild-type or mutated c-kit. Exp Hematol. 2003 Aug;31(8):686-92. doi: 10.1016/s0301-472x(03)00112-7. PMID 12901973
- [Background] Zhang LY, Smith ML, Schultheis B, Fitzgibbon J, Lister TA, Melo JV, Cross NC, Cavenagh JD. A novel K509I mutation of KIT identified in familial mastocytosis-in vitro and in vivo responsiveness to imatinib therapy. Leuk Res. 2006 Apr;30(4):373-8. doi: 10.1016/j.leukres.2005.08.015. Epub 2005 Sep 22. PMID 16183119
- [Background] Ma Y, Zeng S, Metcalfe DD, Akin C, Dimitrijevic S, Butterfield JH, McMahon G, Longley BJ. The c-KIT mutation causing human mastocytosis is resistant to STI571 and other KIT kinase inhibitors; kinases with enzymatic site mutations show different inhibitor sensitivity profiles than wild-type kinases and those with regulatory-type mutations. Blood. 2002 Mar 1;99(5):1741-4. doi: 10.1182/blood.v99.5.1741. PMID 11861291
- [Background] Garcia-Montero AC, Jara-Acevedo M, Teodosio C, Sanchez ML, Nunez R, Prados A, Aldanondo I, Sanchez L, Dominguez M, Botana LM, Sanchez-Jimenez F, Sotlar K, Almeida J, Escribano L, Orfao A. KIT mutation in mast cells and other bone marrow hematopoietic cell lineages in systemic mast cell disorders: a prospective study of the Spanish Network on Mastocytosis (REMA) in a series of 113 patients. Blood. 2006 Oct 1;108(7):2366-72. doi: 10.1182/blood-2006-04-015545. Epub 2006 Jun 1. PMID 16741248
- [Result] Akin C, Fumo G, Yavuz AS, Lipsky PE, Neckers L, Metcalfe DD. A novel form of mastocytosis associated with a transmembrane c-kit mutation and response to imatinib. Blood. 2004 Apr 15;103(8):3222-5. doi: 10.1182/blood-2003-11-3816. Epub 2003 Dec 24. PMID 15070706
- [Result] Hoffmann KM, Moser A, Lohse P, Winkler A, Binder B, Sovinz P, Lackner H, Schwinger W, Benesch M, Urban C. Successful treatment of progressive cutaneous mastocytosis with imatinib in a 2-year-old boy carrying a somatic KIT mutation. Blood. 2008 Sep 1;112(5):1655-7. doi: 10.1182/blood-2008-03-147785. Epub 2008 Jun 20. PMID 18567837